CLINICAL TRIAL: NCT02722876
Title: The EFficacy of COntralateral Muscle Rehabilitation Exercise Following Anterior Cruciate Ligament Reconstruction (EFCOR)
Brief Title: The Efficacy of Rehabilitation Exercise on the Non-operative Limb Following Anterior Cruciate Ligament Reconstruction
Acronym: EFCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: EFCOR001
Record Dates: First submitted 2016-03-17; First posted 2016-03-30 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Musculoskeletal System
Keywords: Rehabilitation; Cross-education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contralateral rehabilitation (Experimental): 8-weeks of resistance training of the non-operative limb following ACL reconstruction
  Interventions: Other: Contralateral Rehabilitation
- Placebo flexibility exercise (Placebo Comparator): 8-weeks of 'placebo' flexibility training of the upper limb
  Interventions: Other: Placebo flexibility exercise

INTERVENTIONS:
Other: Contralateral Rehabilitation — Patients will undergo resistance training of the thigh musculature of the non-injured (contralateral) limb 3 times per week. The exercises will consist of unilateral: knee extensions; knee flexions and; leg-press, all performed on commercially-available resistance training machines. To optimise strength gains, patients will work to the 5 repetition-maximum rule (Kraemer et al. 2002); 3 sets of each exercise will be performed and a 2-minute rest will separate each set. Sessions will take no longer than 15-20 minutes, including rest.
  Arms: Contralateral rehabilitation
Other: Placebo flexibility exercise — Patients will perform 'placebo' flexibility training of the upper limb, which will involve a time-matched stretching programme targeting the latissimus dorsi, triceps brachii, biceps brachii, trapezius and pectoral muscles of both limbs. Each stretch will be performed twice, held for 20-30 seconds each time and will be followed by a 30-second rest (McCrary et al. 2015)
  Arms: Placebo flexibility exercise

SUMMARY:
The purpose of this study is to evaluate the efficacy of a cross-education rehabilitation intervention following anterior cruciate ligament reconstruction on ameliorating the acute losses to function and performance. The cross-education phenomenon describes the strength gain in the opposite, untrained (surgical) limb following unilateral resistance training of the 'trained' (non-surgical) limb.

DETAILED DESCRIPTION:
Protocol:

44 eligible and consenting patients (allowing for 20% attrition) with unilateral anterior cruciate ligament (ACL) injury that have elected to undergo surgical reconstruction will be recruited into this study. Patients will be randomly assigned to one of two different conditions: 1) standard ACL rehabilitation plus 8-weeks of contralateral muscle resistance training, [INTERVENTION]; 2) standard ACL rehabilitation plus placebo exercises (time-matched unrelated upper limb flexibility exercises, [CONTROL].

Assessments of knee extensor and knee flexor neuromuscular performance of both limbs will be obtained prior to, at 10-weeks post- and at 6-months post- surgery. Assessments of function (1-leg hop for distance) and patient-reported outcomes (International Knee Documentation Committee [IKDC]) will also be conducted at these times. Further, all patients will be asked to wear a tri-axial accelerometer to gain an objective measure of habitual physical activity (PA) and sedentary time and pattern for one week pre-surgery (5 weekdays and 2 weekend days), during the first and final week of the INTERVENTION/CONTROL and then again at 6 months post- INTERVENTION/CONTROL.

The initial assessments at 10-weeks post-surgery will evaluate the efficacy of the contralateral training programme, specifically whether the training intervention on the non-injured leg elicited changes in the performance of the injured leg compared to the control group. The assessments at 6-months post-surgery will evaluate any carry-over effects of the contralateral training programme, specifically whether any changes in performance of the injured leg were retained at 6-months post-surgery compared to the control group. 6-months post-surgery is currently the earliest opportunity when we would permit patients to return to sports and activities.

ACL surgeries will be performed by the same three surgeons at the RJAH Orthopaedic Hospital throughout the study and according to standardised techniques and procedures.

Sample size and data analysis:

The means and standard deviations of the primary outcome measure (peak strength) and the correlation coefficient between baseline strength and 8-weeks of strength training, all needed to calculate the sample size, were based on previously accrued data from our laboratory on similar cohorts of ACL patients. Assuming the trial will be powered to detect a difference between the groups of 50N (12.5% of peak strength) with 80% at a two-sided p=0.05 significance level, the trial will require 18 patients in each group assuming analysis will be by ANCOVA (Analysis of Covariance; see formula in Borm et al., 2007). Based on a drop-out rate of 20%, the trial will require a sample size of 22 patients per trial arm (44 patients in total).

Patient recruitment Potential participants will be identified from records of patients listed for ACL surgery and during out-patient clinics. They will be approached by a member of the clinical trial team (consultants, registrars, physiotherapist, lead researcher). The study information and design will be explained to the patients meeting the inclusion criteria and who are interested. They will be given a patient information leaflet and informed consent form to take away with them. These patients will be contacted by phone by the physiotherapist or lead researcher at least 24-hours later to ascertain their verbal consent into the study and to arrange an appointment for an initial assessment. Patients will have the opportunity to ask any questions about the study at this stage also. Written informed consent will be obtained at the first appointment, prior to the initial assessment. Once consented in to the study, patients will be assigned a number. A master copy of individuals' unique identification number and all data will be held on a password-protected computer, stored in a locked cabinet, in a locked NHS research office.

Data monitoring:

Scheduled monthly meetings with the research team will enable monitoring of study progress. Quarterly meetings of the RJAH data monitoring group will provide independent monitoring of the study. No adverse advents are expected, however, ant will be recorded in the on-site file and reported immediately to the data monitoring group.

ELIGIBILITY:
Inclusion Criteria:

* Mentally mature
* Listed for unilateral ACL reconstructive surgery following informed surgical consent
* Autologous graft tissue; either patella tendon or semitendinosus and gracilis from the ipsilateral leg

Exclusion Criteria:

* Patients under 16 or over 50 years of age
* Patients with systemic pathologies (e.g. renal failure)
* Symptomatic non-operative knee
* Additional ligament injuries, meniscal transplant and,or, articular cartilage repair to the operative knee

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Muscle Strength (peak force) | 10-weeks post ACL-reconstruction

SECONDARY OUTCOMES:
Muscle Strength (peak force) | 6-months post ACL-reconstruction
Functional capability | 6-months post ACL-reconstruction
  1-legged hop for distance
Limb symmetry index | 10-weeks and 6-months post ACL-reconstruction
  difference in muscle function between limbs
Patient perceived knee function | 10-weeks and 6-months post ACL-reconstruction
  IKDC questionnaire
Physical activity (PA) | 10-weeks and 6-months post ACL-reconstruction
  Objective measures of PA by accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bailey, PhD, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS FT, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared

REFERENCES:
- [Derived] Minshull C, Gallacher P, Roberts S, Barnett A, Kuiper JH, Bailey A. Contralateral strength training attenuates muscle performance loss following anterior cruciate ligament (ACL) reconstruction: a randomised-controlled trial. Eur J Appl Physiol. 2021 Dec;121(12):3551-3559. doi: 10.1007/s00421-021-04812-3. Epub 2021 Sep 20. PMID 34542671